CLINICAL TRIAL: NCT04859855
Title: Transfusional Trigger in Post-operative Oncologic Patients in Critical Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2789/19
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Transfusion; Oncology; Critical Care; Surgery
Keywords: transfusion; trigger; oncology; post operative; critical care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Transfusion of RBCs according to allocation in two arms: Restrictive strategy (arm A): transfusion if Hb ≤7,0g/dL with the aim of maintaining Hb levels between 7,0-9,0g/dL. Liberal strategy (arm B): transfusion if Hb≤9,0g/dL, with the aim of maintaining Hb levels between 9,0-10,0g/dL. In both arms patients should receive one unit of RBC per time, and Hb should be monitored after 3 hours to check for the need of additional transfusion.
  The strategy should be maintained during the entire ICU stay, for a maximum of 90 days. In case of permanence in the ICU for a period longer than 90 days or if the patient is discharged from the ICU, the transfusional support will be determined by the assisting physicians, independently of the study. If the patient returns to the ICU during the 90 days of randomization, then he should go back to receiving transfusions according to the liberal or restrictive strategy in use previously. Patients will receive pre-storage leukodepleted and irradiated RBCs.
Who Masked: Outcomes Assessor
Masking Description: It will not be feasible to mask the assigned transfusion strategy from health care providers. Information regarding frequency of outcome measures will not be available to the study investigators or health care providers, to minimize comparison of outcomes between study groups. Trial statistician will be blinded for the allocation during analysis. The members of the DMSC will remain blinded unless they request otherwise after the interim analysis provides strong indications of one intervention being beneficial or harmful.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive strategy (arm A) (Experimental): Transfusion of RBC if Hb ≤7,0g/dL with the aim of maintaining Hb levels between 7,0-9,0g/dL.
  Interventions: Procedure: Restrictive transfusional strategy
- Liberal strategy (arm B) (Experimental): Transfusion of RBC if Hb ≤9,0g/dL, with the aim of maintaining Hb levels between 9,0-10,0g/dL.
  Interventions: Procedure: Liberal transfusional strategy

INTERVENTIONS:
Procedure: Restrictive transfusional strategy — Transfusion of Red Blood Concentrates (RBCs) if Hb ≤7,0g/dL with the aim of maintaining Hb levels between 7,0-9,0g/dL.
  Arms: Restrictive strategy (arm A)
Procedure: Liberal transfusional strategy — Transfusion of RBC if Hb ≤9,0g/dL, with the aim of maintaining Hb levels between 9,0-10,0g/dL
  Arms: Liberal strategy (arm B)

SUMMARY:
Transfusional practices evolved significantly over the last decades, but there are still important controversies regarding triggers that should be adopted in different clinical scenarios. Most international guidelines recommend using a hemoglobin (Hb) level around 7,0-8,0g/dL as the value to prompt a transfusion of red blood cell concentrates (RBC). Critical care patients usually are in a hyperdynamic state, working with an elevated cardiac output and compromised organ function. In these patients, the dependency on the arterial content of oxygen is greater, making lower Hb levels more associated with organ disfunction and compromised homeostasis.

With this study the investigators hope to help clinicians to make decisions regarding transfusion of RBCs in critical surgical patients, establishing a transfusional trigger, without exposing patients to unnecessary additional risks, in the scenario involving patients with cancer, in post-operative care.

This is a prospective, randomized, controlled, interventional trial, with the aim of evaluating the impact of restrictive versus liberal transfusional strategy on mortality and severe clinical complications in post-operative oncologic critically ill patients. The primary outcome is mortality in 30 days. The interventions consist in transfusion of RBCs according to the allocation to a liberal or restrictive transfusional strategy. In the restrictive strategy arm patients will receive transfusion of RBCs if the Hb falls to a level equal to or below 7,0g/dL. In the liberal strategy arm patients will receive transfusions if Hb level is below or equal to 9,0g/dL. In both arms patients should receive only one unit of RBC per time, with measurement of Hb level after three hours to evaluate the need for additional units. The strategy should be maintained during intensive care unit (ICU) stay for a maximum of 90 days. In case of a permanence in the ICU for a period longer than 90 days, or if the patient is discharged from the ICU, the transfusional support will be determined by the assisting physicians, independently of the allocated study arm. If the patient returns to the ICU during the 90 days of randomization, then he should go back to receiving transfusions according to the liberal or restrictive strategy in use previously in the ICU.

DETAILED DESCRIPTION:
Randomization: patients will be randomized in a 1:1 ratio to one of the transfusion strategies, stratified according to age ≤65 years or > 65 years.

Monitoring and follow-up: Study investigators will collect all of the necessary data with the use of specific forms during patient study follow up. In case of transfusional reactions related to the RBC transfusions the ICU team should contact the study investigators to notify the reaction. In cases where the termination of participation in the study occurs before completion of 90 days since randomization, a study investigator will contact the patient for collection of information of the final follow-up form. An independent data and safety monitoring committee (DMSC) will review study data every 6 months to check for the need for suspending or terminating the study.

Blinding: It will not be feasible to mask the assigned transfusion strategy from health care providers. Information regarding frequency of outcome measures will not be available to the study investigators or health care providers, to minimize comparison of outcomes between study groups. Trial statistician will be blinded for the allocation during analysis. The members of the DMSC will remain blinded unless otherwise requested after the interim analysis provides strong indications of one intervention being beneficial or harmful.

Interim analysis: an interim analysis will be performed when a total of 420 patients (half of the expected target sample) has completed 90 days of follow-up. The independent DMSC will recommend interruption of the trial if the difference in the primary outcome measure between groups has a P <0.001 (Haybittle-Peto criterion).

The trial protocol may be temporarily suspended for an individual patient in case of arterial ischemic events (includes stroke, myocardial infarction, unstable angina, mesenteric ischemia, peripheral ischemia) or life-threatening bleeding, at the discretion of the attending physician. The patient may re-enter the trial protocol after stabilization, at the discretion of the attending doctor.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a solid tumor and age ≥ 18 years
* Admission to the ICU due to postoperative care after being submitted to a major surgical procedure (defined as having a duration of three hours or more)
* Expected ICU stay of more than 24 hours
* Presenting Hb value of 9,0g/dL or less during ICU stay, within the first 7 days post-surgical procedure

Exclusion Criteria:

* Hematological malignancy
* Chronic anemia (defined as presenting Hb ≤9,0g/dL at hospital admission and / or diagnosed hematological disease)
* Presence of active bleeding at the moment of inclusion in the study (defined as visible bleeding with fall of 2,0g/dL in Hb levels in the last 12 hours or need to reoperate)
* Transfusion of RBC during the current ICU stay before the inclusion in the study
* Patient refusal to receive blood transfusions
* Pregnancy
* Postoperative care of cardiac surgery or surgery for correction of hip fracture
* Patients with terminal oncological disease in palliative care
* Arterial ischemic event in the current hospital stay or in the past twelve months (includes stroke, myocardial infarction, unstable angina, mesenteric ischemia, peripheral ischemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality | 30 days
  Mortality 30 days post-randomization

SECONDARY OUTCOMES:
Rate of mortality at 60 and 90 days post-randomization | 60 and 90 days
  Mortality at 60 and 90 days post-randomization
Rate of mortality in hospital and ICU admission | 90 days after randomization
  Mortality in hospital and ICU admission
Number of days alive | 90 days after randomization
  Days alive during the 90 days after randomization
Duration of ICU and hospital stay | 90 days after randomization
  Duration of ICU and hospital stay
Number of days alive and out of the hospital during the 90 days after randomization | 90 days after randomization
  Days alive and out of the hospital during the 90 days after randomization
Rate of organ dysfunction | 90 days after randomization
  Total frequency of events: acute renal failure requiring dialysis, acute respiratory distress syndrome with need of mechanical ventilation, hemodynamic instability with need of vasopressor/inotropic therapy, congestive heart failure
Number of days alive without mechanical ventilation | 90 days after randomization
  Days alive without mechanical ventilation 90 days after randomization
Number of days alive without vasopressor/inotropic therapy | 90 days after randomization
  Days alive without vasopressor/inotropic therapy 90 days after randomization
Number of days alive without dialysis/hemofiltration 90 days after randomization | 90 days after randomization
  Days alive without dialysis/hemofiltration
Rate of acute ischemic events occurring in the ICU | 90 days after randomization
  Total frequency of events: stroke, myocardial infarction, unstable angina, mesenteric ischemia, peripheral ischemia
Total frequency of verified infections during ICU admission | 90 days after randomization
  Total frequency of verified infections during ICU admission
Rate of severe adverse transfusional reactions | 90 days after randomization
  Total frequency of events: severe anaphylactic/allergic reactions, acute hemolysis, transfusion-associated lung injury (TRALI), transfusion associated circulatory overload (TACO)
Rate of reoperation | 90 days after randomization
  Not previously programmed

CONTACTS AND LOCATIONS:
Overall Officials: Marina P Colella, MD PhD, Principal Investigator — ACCamargo Cancer Center/ State University of Campinas
Locations (1):
- ACCamargoCC, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Carson JL, Duff A, Poses RM, Berlin JA, Spence RK, Trout R, Noveck H, Strom BL. Effect of anaemia and cardiovascular disease on surgical mortality and morbidity. Lancet. 1996 Oct 19;348(9034):1055-60. doi: 10.1016/S0140-6736(96)04330-9. PMID 8874456
- [Background] Carson JL, Noveck H, Berlin JA, Gould SA. Mortality and morbidity in patients with very low postoperative Hb levels who decline blood transfusion. Transfusion. 2002 Jul;42(7):812-8. doi: 10.1046/j.1537-2995.2002.00123.x. PMID 12375651
- [Background] Carson JL, Stanworth SJ, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2016 Oct 12;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub4. PMID 27731885
- [Background] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Background] de Almeida JP, Vincent JL, Galas FR, de Almeida EP, Fukushima JT, Osawa EA, Bergamin F, Park CL, Nakamura RE, Fonseca SM, Cutait G, Alves JI, Bazan M, Vieira S, Sandrini AC, Palomba H, Ribeiro U Jr, Crippa A, Dalloglio M, Diz Mdel P, Kalil Filho R, Auler JO Jr, Rhodes A, Hajjar LA. Transfusion requirements in surgical oncology patients: a prospective, randomized controlled trial. Anesthesiology. 2015 Jan;122(1):29-38. doi: 10.1097/ALN.0000000000000511. PMID 25401417
- [Background] Holst LB, Haase N, Wetterslev J, Wernerman J, Guttormsen AB, Karlsson S, Johansson PI, Aneman A, Vang ML, Winding R, Nebrich L, Nibro HL, Rasmussen BS, Lauridsen JR, Nielsen JS, Oldner A, Pettila V, Cronhjort MB, Andersen LH, Pedersen UG, Reiter N, Wiis J, White JO, Russell L, Thornberg KJ, Hjortrup PB, Muller RG, Moller MH, Steensen M, Tjader I, Kilsand K, Odeberg-Wernerman S, Sjobo B, Bundgaard H, Thyo MA, Lodahl D, Maerkedahl R, Albeck C, Illum D, Kruse M, Winkel P, Perner A; TRISS Trial Group; Scandinavian Critical Care Trials Group. Lower versus higher hemoglobin threshold for transfusion in septic shock. N Engl J Med. 2014 Oct 9;371(15):1381-91. doi: 10.1056/NEJMoa1406617. Epub 2014 Oct 1. PMID 25270275
- [Background] Hovaguimian F, Myles PS. Restrictive versus Liberal Transfusion Strategy in the Perioperative and Acute Care Settings: A Context-specific Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesthesiology. 2016 Jul;125(1):46-61. doi: 10.1097/ALN.0000000000001162. PMID 27167445
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Hebert PC, Yetisir E, Martin C, Blajchman MA, Wells G, Marshall J, Tweeddale M, Pagliarello G, Schweitzer I; Transfusion Requirements in Critical Care Investigators for the Canadian Critical Care Trials Group. Is a low transfusion threshold safe in critically ill patients with cardiovascular diseases? Crit Care Med. 2001 Feb;29(2):227-34. doi: 10.1097/00003246-200102000-00001. PMID 11246298
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Management. Practice guidelines for perioperative blood management: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Management*. Anesthesiology. 2015 Feb;122(2):241-75. doi: 10.1097/ALN.0000000000000463. No abstract available. PMID 25545654
- [Background] Shander A, Javidroozi M, Naqvi S, Aregbeyen O, Caylan M, Demir S, Juhl A. An update on mortality and morbidity in patients with very low postoperative hemoglobin levels who decline blood transfusion (CME). Transfusion. 2014 Oct;54(10 Pt 2):2688-95; quiz 2687. doi: 10.1111/trf.12565. Epub 2014 Feb 17. PMID 24527739
- [Background] Taira R, Satake M, Momose S, Hino S, Suzuki Y, Murokawa H, Uchida S, Tadokoro K. Residual risk of transfusion-transmitted hepatitis B virus (HBV) infection caused by blood components derived from donors with occult HBV infection in Japan. Transfusion. 2013 Jul;53(7):1393-404. doi: 10.1111/j.1537-2995.2012.03909.x. Epub 2012 Oct 4. PMID 23033944
- [Background] Vieira PCM, Lamarao LM, Amaral CEM, Correa ASM, de Lima MSM, Barile KADS, de Almeida KLD, Sortica VA, Kayath AS, Burbano RMR. Residual risk of transmission of human immunodeficiency virus and hepatitis C virus infections by blood transfusion in northern Brazil. Transfusion. 2017 Aug;57(8):1968-1976. doi: 10.1111/trf.14146. Epub 2017 Jun 7. PMID 28589643
- [Background] Wang JK, Klein HG. Red blood cell transfusion in the treatment and management of anaemia: the search for the elusive transfusion trigger. Vox Sang. 2010 Jan;98(1):2-11. doi: 10.1111/j.1423-0410.2009.01223.x. Epub 2009 Aug 4. PMID 19682346
- [Background] Weiskopf RB, Feiner J, Hopf H, Viele MK, Watson JJ, Lieberman J, Kelley S, Toy P. Heart rate increases linearly in response to acute isovolemic anemia. Transfusion. 2003 Feb;43(2):235-40. doi: 10.1046/j.1537-2995.2003.00302.x. PMID 12559019
- [Background] Weiskopf RB, Viele MK, Feiner J, Kelley S, Lieberman J, Noorani M, Leung JM, Fisher DM, Murray WR, Toy P, Moore MA. Human cardiovascular and metabolic response to acute, severe isovolemic anemia. JAMA. 1998 Jan 21;279(3):217-21. doi: 10.1001/jama.279.3.217. PMID 9438742
- [Background] Wu WC, Schifftner TL, Henderson WG, Eaton CB, Poses RM, Uttley G, Sharma SC, Vezeridis M, Khuri SF, Friedmann PD. Preoperative hematocrit levels and postoperative outcomes in older patients undergoing noncardiac surgery. JAMA. 2007 Jun 13;297(22):2481-8. doi: 10.1001/jama.297.22.2481. PMID 17565082
- [Background] Fossaluza V, Diniz JB, Pereira Bde B, Miguel EC, Pereira CA. Sequential allocation to balance prognostic factors in a psychiatric clinical trial. Clinics (Sao Paulo). 2009;64(6):511-8. doi: 10.1590/s1807-59322009000600005. PMID 19578654